CLINICAL TRIAL: NCT01778933
Title: A Pilot and Feasibility Study Of The Imaging Potential Of EC17 In Subjects Undergoing Surgery Presenting With Renal Nodules
Brief Title: Intraoperative Imagery of Renal Nodules With Folate-fluorescein Conjugate(EC17)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sunil Singhall, Assistant Professor of Medicine, Assistant Professor of Surgery, Director Thoracic Surgery Research Laboratory, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC17 Renal Cell; 816726 (Other: UPenn IRB Protocol #)
Record Dates: First submitted 2013-01-18; First posted 2013-01-29 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-03

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal cell carcinoma; Renal nodules
MeSH Terms: conditions — Carcinoma, Renal Cell

ARMS (1):
- EC17 Injection Group (Experimental): The group will receive a single dose of EC17, infused over 10 minutes, prior to surgery. Then, during surgery, the EC-17 will be imaged with a camera that the investigators have developed.
  Interventions: Drug: EC17

INTERVENTIONS:
Drug: EC17

SUMMARY:
According to the National Cancer Institute, an estimated 64,770 men and women will be diagnosed with kidney cancer in 2012. Of this number, an estimated 13,570 will die of this disease. Surgery remains one of the best options for patients presenting with operable Stage II or III cancers, however the five year survival rate for these candidates remains at a dismal 63.7% for Stage II and 11% for Stage III. The high rates of recurrence suggest that surgeons are unable to completely detect and remove primary tumor nodules in a satisfactory manner as well as lingering metastases in sentinel lymph nodes. By ensuring a negative margin through imaging during surgery it would be possible for the investigators to improve the rates of recurrence free patients and thus overall survival.

Renal cell malignancies are the ideal disease to investigate intra-operative imaging. 70% of kidney malignancies express folate receptor alpha (FRA). It is important to note that FRA is expressed only in the proximal tubules of the kidneys, activated macrophages, and in the choroidal plexus. Thus, the false positive detection rate is expected to be extremely low. A group well known to us in the Netherlands has completed a pilot study utilizing a folate-FITC conjugate in 12 patients with ovarian cancer. Another group of investigators in Mayo have subsequently performed this study on 20 more patients without any serious adverse events (personal communication). They report excellent sensitivity and specificity with this technique with only grade 1 side effects (allergic reaction). All side effects reversed when the injection was halted. Patients with a history of allergic reactions to insect bites should not participate (fluorescein is derived from the firefly insect, folate is an essential vitamin).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years of age or older
2. Patients presenting with a renal cell nodule or mass that are scheduled for open or laparoscopic resection based on clinical criteria
3. Good operative candidate
4. Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria:

1. Pregnant women as determined by urinary or serum beta human chorionic gonadotropin (hCG) test within 72 hours of surgery
2. Patients with a history of anaphylactic reactions to Folate-FITC or insects
3. At-risk patient populations

   1. People who would be easily lost to follow-up (ex: People who are homeless or alcohol dependent)
   2. Children and neonates
   3. Patients unable to participate in the consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The ability of EC17 and the imaging system to detect FRA positive tumors during surgery conducted 2-4 hours post EC-17 administration. | Within two to four hours of injection of the EC17

SECONDARY OUTCOMES:
The number of participants that will have an adverse reaction to the EC17 | Day 1 - Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Guzzo TJ, Jiang J, Keating J, DeJesus E, Judy R, Nie S, Low P, Lal P, Singhal S. Intraoperative Molecular Diagnostic Imaging Can Identify Renal Cell Carcinoma. J Urol. 2016 Mar;195(3):748-55. doi: 10.1016/j.juro.2015.09.093. Epub 2015 Nov 2. PMID 26541080